CLINICAL TRIAL: NCT07391969
Title: Evaluation of New Supraglottic Airway Device - SaCo VLMA for General Anesthesia for Laparoscopic Procedures
Brief Title: Evaluation of SaCo VLMA for General Anesthesia for Laparoscopic Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Gaszynski, prof. dr hab., Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RNN/120/23/KE
Record Dates: First submitted 2026-01-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Laparoscopic Surgical Procedures; Airway Control; Anesthesia
MeSH Terms: interventions — Sagittal Abdominal Diameter; Airway Management; Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the collected data will be anonymized regarding used for airway control device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaCo VLMA airway management (Experimental): SaCo VLMA Supraglottic Airway Device for airway control in anesthetized patient for general anesthesia for laparoscopic surgery
  Interventions: Device: SaCo VLM or SAD or ET for airway control for laparoscopy
- Other device for airway management (Active Comparator): Other Airway Device for airway control in anesthetized patient for general anesthesia for laparoscopic surgery
  Interventions: Device: SaCo VLM or SAD or ET for airway control for laparoscopy

INTERVENTIONS:
Device: SaCo VLM or SAD or ET for airway control for laparoscopy — Evaluation of the new SGAs for airway control in anesthetized patients for laparoscopy procedures

SUMMARY:
Evaluation of new supraglottic device SaCo VLMA for laparoscopic procedures under general anesthesia in comparison with other airway management methods including other supraglottic devices. The parameters noted will be: demographic data, time for placement of SGA counted from moment of grabbing device by operator to correct placement, subjective evaluation of ease of insertion of SGA in 5 step Borg scale, peak pressure, lung compliance, achieved tidal volume before creating pneumoperitoneum, after creating pneumoperitoneum, visualization of glottis on monitor of camera or fiberoptic scope.

DETAILED DESCRIPTION:
Evaluation of new supraglottic device SaCo VLMA for laparoscopic procedures under general anesthesia in comparison of other supraglottic devices and other methods of airway management for such procedures.

The airway management for laparoscopic surgery can be achieved by either endotracheal intubation (ET) or use of supraglottic devices (SGA). However, many anesthesiologist still prefer ET over use of SGA because of possible problems with adequate ventilation during pneumoperitoneum.

New SGA devices as video laryngeal mask offer important advantage which is continuous control of proper placement of SGA during anesthesia. In case of ventilation difficulties like leak, high peak pressure, low tidal volume SGA VLM allow to check if the problem is related to malposition or changed of position of SGA and allow for correction under control of vision.

The aim of this study is to evaluate the characteristics of the SaCo VLMA video laryngeal mask in the hands of experienced anesthesiologists.

All patients will be anesthetized following the same protocol: Intravenous induction with propofol, FNT, midazolam, rocuronium in standard doses. After achieving proper muscle relaxation SaCo VLMA was inserted following manufacturer recommendations. For maintaining anesthesia sevoflurane was used.

After induction for anesthesia the airway of the patient will be secured by one randomly chosen device: SaCo VLMA or other SGA or ET.

The parameters noted will be: demographic data, time for placement of SGA counted from moment of grabbing device by operator to correct placement, subjective evaluation of ease of insertion of SGA in 5 step Borg scale, peak pressure, lung compliance, achieved tidal volume before creating pneumoperitoneum, after creating pneumoperitoneum, visualization of glottis on monitor of camera or fiberoptic scope.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery under general anesthesia for laparoscopic surgery of predicting lasting no longer than about 1 hour.
* Age >18 years.
* ASA I-III.
* Present ordinary airway

Exclusion Criteria:

* Not meeting the above criteria
* Presenting 3 predictors of a difficult airway (Mallampatti class III or IV; thyromental distance <6 cm, sternomental distance <12.5 cm, distance between incisors <4.0 cm, bite test II or III, cervical mobility <90o).
* Gestation
* Allergy to any drug included in the protocol.
* Present risk factors for bronchial aspiration

  - Presenting with preoperative sore throat
* Present severe respiratory, coronary or cerebral vascular pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
effectiveness of use | immediately after the intervention
  success ratio of insertion of SGA or ET in % of success insertion
effectiveness of mechanical ventilation | perioperatively
  adequate ventilation described as maintaining adequate minute ventilation with acceptable leak in Tidal Volume in ml
safety of mechanical ventilation | perioperatively
  providing adequate ventilation parameters - peak pressure in mmHg
parameters of mechanical ventilation | perioperatively
  measurement of lung compliance in ml/mmHg

SECONDARY OUTCOMES:
safety of use of SaCo VLM | immediately after the surgery
  complications ratio related to airway management in %

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Principal Investigator — Medical University of Lodz

IPD SHARING:
Plan to Share IPD: No